CLINICAL TRIAL: NCT00933140
Title: Anal HPV Infection and Abnormal Cytology in HIV-infected Women
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Stier, Attending and Associate Professor, Boston Medical Center
Other Study IDs: H-25758
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Cervical Cancer Screening; HIV Infections
Keywords: HIV; women; anal cytology
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV infected women: HIV infected women between ages 18 - 64 years of age due for cervical cancer screening were enrolled.

SUMMARY:
The population of HIV infected women seen at Boston Medical Center may have a higher frequency of anal cytologic and histologic abnormalities than what is reported for the non-HIV infected population.

DETAILED DESCRIPTION:
BACKROUND FOR THIS STUDY Anal cancer is a growing problem in the US. The incidence of anal cancer has increased among both men (160%) and women (78%) from 1973 to 2000 in the US [1]. In HIV-infected men the incidence of SCCA (squamous cell cancer of the anus) was found to range from 49-92 per 100,000 patient years [2]. This prompted recommendations on screening for anal cancer in this population. HIV-infected women are also at increased risk for developing anal cancer. A study based on data from AIDS and cancer registries found that the risk of anal cancer among women in the general population is about 1.2% and it increases up to 3.9% in the HIV-infected women. In addition, HIV-infected women had eight times the risk of in situ anal cancer compared with the number of expected cases [3].

SCCA appears to have many similarities to cervical cancers. HPV has been detected in 88% of anal cancer specimens with HPV-16 found in 73% of SCCA and HPV-18 in 7% [1]. In addition, SCCA develops in the transformation zone between the squamous epithelium of the anus and the columnar epithelium of the rectum, is frequently associated with dysplasia of the anus and may be preceded by squamous intraepithelial changes which are also associated with HPV.

Cervical cytology, also known as pap smear, can detect cervical cancer and its precursors. Countries who have adopted cervical cancer screening programs have had dramatic decreases in both the morbidity and mortality rates of cervical cancer.

Anal cytology may also be used to screen for HPV associated anal lesions, and among HIV-infected men who have sex with men, an abnormal cytology is frequently associated with a dysplastic squamous cell lesion of the anus. Anal HPV infections (high risk types) have been found in 53 ¿ 95% of HIV-infected men. Abnormal anal cytology has been found in 41-81% of HIV-infected men screened with high-grade cytologic findings in 2-25% of these patients [2].

There have been only a few studies looking at anal cytology in HIV-infected women. The largest study (n=235), by Holly and Palefsky [4], found that HIV positive women had a 26% prevalence of anal cytologic abnormalities (mostly atypical squamous cells of undetermined significance [ASCUS] and low grade squamous intraepithelial lesions [LSIL]). Forty-six of these women with abnormal cytology (60) underwent high resolution anoscopy (HRA) and 14 were found to have biopsy proven HSIL.

Several risk factors for anal cytologic abnormalities in women have been suggested, such as positive anal HPV test, history of anal intercourse, history of cervical squamous intraepithelial lesions (SIL), history of vulvar warts, multifocal cervical SIL, history of sexually transmitted infections, more than 10 sexual partners, history of cervical, vulvar or vaginal cancer, immunosuppression after solid organ transplantation, HIV infection, long-term corticosteroids use and cigarette smoking.

It has been suggested that all HIV-infected women, women with cervical cancer and women with high-grade vulvar disease or cancer should be screened for anal cytologic abnormalities. However, as described above there is very scanty literature describing the prevalence and incidence in this patient population and the largest study was conducted prior to the HAART era.

We plan to estimate the prevalence and 6-12 month incidence of abnormal anal cytology with histologic correlates in the HIV-infected women seen at BMC. We hope that the information will allow us to make screening recommendations for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64 years
* HIV infected women
* due for cervical cytologic screening

Exclusion Criteria:

* Pregnancy
* On chronic anticoagulation medication
* Life expectancy of the woman is less than 1 year
* If the woman has had a cervical or anal pap test in the last 6 months

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV infected women aged between 18-64 years presenting for cervical cytologic screening.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Primary objective is to determine the rate of anal cytologic and histologic abnormalities in HIV infected women at Boston Medical Center. | 2 years

SECONDARY OUTCOMES:
Identify risk factors for anal cytologic and histologic abnormalities in HIV infected women at BMC | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Stier, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States